CLINICAL TRIAL: NCT05142982
Title: FDG PET-CT Based Risk Adapted Radiotherapy vs Observation for Post Chemotherapy Residual Mass in Advanced Seminoma: A Prospective Randomised Controlled Trial
Brief Title: Radiotherapy vs Observation for Post Chemotherapy Residual Mass in Advanced Seminoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Vedang Murthy, Professor, Tata Memorial Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROsem
Record Dates: First submitted 2021-11-15; First posted 2021-12-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Seminoma
Keywords: FDG-PET CT, radiotherapy
MeSH Terms: conditions — Seminoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy (Experimental): Patients randomized to the test arm will undergo radiotherapy to the residual mass. Patients will be stratified by the size of the residual mass in shortest dimension being <3 cm or > 3 cm.A dose of 30-36 Gy in conventional fractionation of 1.8-2.0 Gy per fraction using 3-dimensional conformal technique. Radiotherapy will be delivered five days a week.
  Interventions: Radiation: Radiotherapy
- Observation (No Intervention): Patients randomized to the standard arm will be observed and the status of residual mass monitored with an FDG PETCT scan done at three to six monthly intervals.

INTERVENTIONS:
Radiation: Radiotherapy — A dose of 30-36 Gy in conventional fractionation of 1.8-2.0 Gy per fraction using 3-dimensional conformal technique. Radiotherapy will be delivered five days a week.
  Arms: Radiotherapy

SUMMARY:
Testicular tumors account for 1% of all cancers in males and germ cell tumors comprise 95% of all testicular cancers. Seminomas consist of around 50% of cases. However,adequate information is not there as 60- 80% residual disease is seen even after with the standard management of chemotherapy.

With the advent of functional imaging there was hope that it could aid in more accurately targeting these tumors to systematically evaluate the role of PET-CT imaging in identifying patients diagnosed with stage IIB-IIIC seminomatous germ cell tumor, with residual visible tumor post chemotherapy who would benefit with loco regional radiotherapy.

The therapeutic research in Seminomashas been relatively slow and such structured studies can allow analysis of large number of patients to report on acute and late effect of treatment outcomes using CTCAE and QOL (EORTC QLQ C-30) in these cancers. We hope that we will get help in identifying thrust areas for future research through this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of classical seminoma
2. Primary site - testis, mediastinum or retroperitoneum
3. Stage IIB-IIIC (AJCC 8th edition)
4. Age>18 years
5. Karnofsky Performance Status at least 70
6. A response assessment FDG PETCT scan done at least twelve weeks after the first line chemotherapy, showing a persistent measurable residual mass
7. Patient willing and reliable for follow up and QOL.

Exclusion Criteria:

1. Histology other than classical seminoma
2. Non completion of planned first-line chemotherapy
3. Prior history of radiotherapy to the involved region
4. Inability to deliver adequate radiotherapy dose safely based on assessment by radiation oncologist

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 2 years
  • Progression free survival (PFS) is defined as the time period from the date of enrolment in the study till the first observation of disease progression at any site, or death.

SECONDARY OUTCOMES:
Locoregional control (LRC) | 2 years
  • Locoregional control (LRC) defined as the time period from the date of enrolment in the study till the first observation of disease progression locally and/or in the regional lymph nodes, or death.
Overall survival (OS) | 2 years
  • Overall survival (OS) defined as the time period from the date of enrolment in the study till the date of death.
Second-line salvage therapy-free survival | 2 years
  • Second-line salvage therapy-free survival defined as the time period from the date of enrolment in the study till date of starting second-line chemotherapy.
Acute radiation toxicity | 2 years
  Incidence of Acute radiation toxicity will be defined as any toxicity within 90 days post RT using RTOG and CTCAE
Late radiation toxicity | 2 years
  Incidence of late radiation toxicity defined as any toxicity after 90 days of post RT using RTOG and CTCAE
Patient-reported quality of life (QOL) | 2 years
  Patient-reported quality of life (QOL) will be assessed using the EORTC QLQ-C30 questionnaire's validated translations in English, Hindi, and Marathi.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Dr Vedang Murthy, Navi Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No